CLINICAL TRIAL: NCT05394792
Title: CANadian Effectiveness of UPadacitinib in Adult Moderate-to-severe aTopIc derMatitis Patients Who Are Inadequate Responders to Dupilumab or diScontinuing Dupilumab Due to safEty/Tolerability Reasons: The CAN UpTIMISE Study
Brief Title: An Observational Study of Upadacitinib to Assess Change in Disease Activity in Canadian Adult Participants With Moderate-to-Severe Atopic Dermatitis Who Are Inadequate Responders To or Discontinuing Dupilumab
Acronym: CAN UpTIMISE
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P23-106
Record Dates: First submitted 2022-05-25; First posted 2022-05-27 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis (AD); Upadacitinib; RINVOQ
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants Receiving Upadacitinib: Participants receiving upadacitinib for moderate to severe atopic dermatitis.

SUMMARY:
Atopic dermatitis (AD) is a skin condition that may cause a rash and itching due to inflammation of the skin. Therapies spread over the skin may not be enough to control the AD in trial participants who require systemic anti-inflammatory treatment. This study will assess the real-world effectiveness of upadacitinib on adult participants with moderate-to-severe AD who are inadequate responders to dupilumab or who are discontinuing from dupilumab due to safety/tolerability reasons. This study also aims to understand upadacitinib utilization patterns in real-world clinical practice.

In Canada, upadacitinib is indicated for the treatment of adults and adolescents 12 years of age and older with refractory moderate to severe atopic dermatitis (AD) who are not adequately controlled with a systemic treatment (e.g., steroid or biologic) or when use of those therapies is inadvisable. CAN UpTIMISE will enroll approximately 100 adult participants, 18 years of age and above, with moderate-to-severe AD who are inadequate responders to dupilumab or are discontinuing from dupilumab from up to 25 sites in Canada.

Participants will receive oral upadacitinib tablets as prescribed by the physician prior to enrolling in this study in accordance with the terms of the local marketing authorization and professional and reimbursement guidelines with regards to dose, population, and indication. The overall duration of the study is approximately 4 Months.

Participants will attend regular visits per routine clinical practice. The effect of the treatment will be checked by medical assessments, using questionnaires, and reporting potential side-effects.

ELIGIBILITY:
Inclusion Criteria:

* Able to give written informed consent before starting any study-related assessments
* Diagnosis of moderate or severe AD, as per investigator's judgement
* Initiating upadacitinib treatment, as per the local label, and where decision to treat with upadacitinib must have been made with the participant, prior to and independently of enrolment in the study
* Previous treatment with dupilumab for AD, as the most recent systemic therapy, and who is either or:

  * i. sub-optimally controlled as per investigator judgement, after at least 16 weeks of dupilumab treatment, with or without additional AD therapies, at time of baseline visit.
  * ii. discontinuing dupilumab due to safety/tolerability reason(s) as per investigator judgement at the baseline visit
* Availability of medication history during the past 4 weeks prior to baseline visit

Exclusion Criteria:

* Previous treatment with any systemic JAKi including upadacitinib, or any investigational drug of chemical or biologic nature within 4 weeks or five half-lives of the drug (whichever is longer) prior to and at the time of the baseline visit
* Currently enrolled in an interventional clinical study, or within the last 30 days or five-half lives of being administered an investigational drug, whichever is longer, prior to baseline visit. Participation in other observational studies or registries is acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with moderate-to-severe Atopic Dermatitis who are inadequate responders to dupilumab or are discontinuing from dupilumab due to safety/tolerability reasons.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Validated Investigator Global Assessment for Atopic Dermatitis (vlGA-AD) of 0 or 1 | Month 4
  vIGA-AD is a validated assessment instrument used in clinical studies to rate the severity of AD globally. A 5-point scale is used to measure the severity of disease at the time of the investigator's evaluation of the participant ranging from 0 - Clear (no inflammatory signs of atopic dermatitis (no erythema, no induration/papulation, no lichenification, no oozing/crusting). Post-inflammatory hyperpigmentation and/or hypopigmentation may be present.) to 4 - Severe (marked erythema (deep or bright red), marked induration/papulation, and/or marked lichenification.

SECONDARY OUTCOMES:
Percentage of Participants Achieving vlGA-AD of 0 or 1 | Up to 2 Months
  vIGA-AD is a validated assessment instrument used in clinical studies to rate the severity of AD globally. A 5-point scale is used to measure the severity of disease at the time of the investigator's evaluation of the participant ranging from 0 - Clear (no inflammatory signs of atopic dermatitis (no erythema, no induration/papulation, no lichenification, no oozing/crusting). Post-inflammatory hyperpigmentation and/or hypopigmentation may be present.) to 4 - Severe (marked erythema (deep or bright red), marked induration/papulation, and/or marked lichenification.
Percentage of Participants Achieving vlGA-AD of ≥ 2 at baseline reaching a vIGA-AD score of 0 or 1 | Up to 4 Months
  vIGA-AD is a validated assessment instrument used in clinical studies to rate the severity of AD globally. A 5-point scale is used to measure the severity of disease at the time of the investigator's evaluation of the participant ranging from 0 - Clear (no inflammatory signs of atopic dermatitis (no erythema, no induration/papulation, no lichenification, no oozing/crusting). Post-inflammatory hyperpigmentation and/or hypopigmentation may be present.) to 4 - Severe (marked erythema (deep or bright red), marked induration/papulation, and/or marked lichenification.
Percentage of Participants with a vIGA score 0 or 1 at Baseline Maintaining a vIGA-AD score 0 or 1 | From Baseline to Month 4
  vIGA-AD is a validated assessment instrument used in clinical studies to rate the severity of AD globally. A 5-point scale is used to measure the severity of disease at the time of the investigator's evaluation of the participant ranging from 0 - Clear (no inflammatory signs of atopic dermatitis (no erythema, no induration/papulation, no lichenification, no oozing/crusting). Post-inflammatory hyperpigmentation and/or hypopigmentation may be present.) to 4 - Severe (marked erythema (deep or bright red), marked induration/papulation, and/or marked lichenification.
Percentage of Participants with an Eczema Area and Severity Index (EASI) score corresponding to, at least, mild disease (≥1.1) at baseline achieving an absolute EASI score corresponding to clear or almost clear disease (<1.1) | Up to 4 Months
  EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
Percentage of Participants with an EASI score corresponding to, at least, moderate disease (≥7.1) at baseline achieving an absolute EASI score corresponding to mild disease (<7.1) | Up to 4 Months
  EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
Absolute mean EASI score | Up to 4 Months
  EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
Percent change in EASI score from baseline | Up to 4 Months
  EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
Mean change in EASI score from baseline | Up to 4 Months
  EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
Percent change in EASI score by body region (head and neck region, trunk [including genitals], upper limbs, and lower limbs [including buttocks]) | Up to 4 Months
  EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
Mean change in EASI score by body region (head and neck region, trunk [including genitals], upper limbs, and lower limbs [including buttocks]) | Up to 4 Months
  EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
Percent change in Worst pruritus numerical rating scale (WP-NRS) score from baseline | Up to 4 Months
  WP-NRS is a validated single self-reported item designed to measure peak pruritus, or 'worst' itch, over the previous 24 hours with a higher score denoting worse itch.
Mean change in WP-NRS score from baseline | Up to 4 Months
  WP-NRS is a validated single self-reported item designed to measure peak pruritus, or 'worst' itch, over the previous 24 hours with a higher score denoting worse itch.
Percentage of Participants with WP-NRS >2 at baseline achieving a WP-NRS score of 0 or 1 | Up to 4 Months
  WP-NRS is a validated single self-reported item designed to measure peak pruritus, or 'worst' itch, over the previous 24 hours with a higher score denoting worse itch.
Percentage of Participants achieving Dermatology Life Quality Index (DLQI) score of 0 or 1 | Up to 4 Months
  DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on health-related quality of life (HRQoL). It consists of 10 questions assessing impact of skin diseases on different aspects of subject's QoL over the prior week. Each item is scored on a 4-point scale: 0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much. Item scores (0 to 3) are added to provide a total score range of 0 to 30. Higher scores indicate greater impairment of HRQoL.
Percentage of Participants with a baseline DLQI score ≥ 2 (at least small effect on participant's quality of life) achieving a DLQI score of 0 or 1 | Up to 4 Months
  DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on health-related quality of life (HRQoL). It consists of 10 questions assessing impact of skin diseases on different aspects of subject's QoL over the prior week. Each item is scored on a 4-point scale: 0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much. Item scores (0 to 3) are added to provide a total score range of 0 to 30. Higher scores indicate greater impairment of HRQoL.
Absolute mean DLQI scores | Up to 4 Months
  DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on health-related quality of life (HRQoL). It consists of 10 questions assessing impact of skin diseases on different aspects of subject's QoL over the prior week. Each item is scored on a 4-point scale: 0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much. Item scores (0 to 3) are added to provide a total score range of 0 to 30. Higher scores indicate greater impairment of HRQoL.
Percent change in DLQI score from Baseline | Up to 4 Months
  DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on health-related quality of life (HRQoL). It consists of 10 questions assessing impact of skin diseases on different aspects of subject's QoL over the prior week. Each item is scored on a 4-point scale: 0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much. Item scores (0 to 3) are added to provide a total score range of 0 to 30. Higher scores indicate greater impairment of HRQoL.
Mean change in DLQI score from Baseline | Up to 4 Months
  DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on health-related quality of life (HRQoL). It consists of 10 questions assessing impact of skin diseases on different aspects of subject's QoL over the prior week. Each item is scored on a 4-point scale: 0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much. Item scores (0 to 3) are added to provide a total score range of 0 to 30. Higher scores indicate greater impairment of HRQoL.
Absolute mean Patient Oriented Eczema Measurement (POEM) score | Up to 4 Months
  The POEM is a 7-item, validated questionnaire used in clinical practice and clinical trials to assess disease symptoms in both children and adults. Participants respond to 7 items, including dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping, each scored on a 5-point scale based on frequency over the previous week: 0 = no days, 1 = 1 to 2 days, 2 = 3 to 4 days, 3 = 5 to 6 days, and 4 = all days. Item scores (0 to 4) are added to provide a total score range of 0 to 28. The total score reflects disease-related morbidity, and differentiates between "clear/almost clear" (0-2 points), "mild" (3-7 points), "moderate" (8-16 points), "severe" (17-24 points) and "very severe" (25-28 points) AD. A change in POEM score of 3.4 points is considered the MCID.
Percent change in POEM score from baseline | Up to 4 Months
  The POEM is a 7-item, validated questionnaire used in clinical practice and clinical trials to assess disease symptoms in both children and adults. Participants respond to 7 items, including dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping, each scored on a 5-point scale based on frequency over the previous week: 0 = no days, 1 = 1 to 2 days, 2 = 3 to 4 days, 3 = 5 to 6 days, and 4 = all days. Item scores (0 to 4) are added to provide a total score range of 0 to 28. The total score reflects disease-related morbidity, and differentiates between "clear/almost clear" (0-2 points), "mild" (3-7 points), "moderate" (8-16 points), "severe" (17-24 points) and "very severe" (25-28 points) AD. A change in POEM score of 3.4 points is considered the MCID.
Mean change in POEM score from baseline | Up to 4 Months
  The POEM is a 7-item, validated questionnaire used in clinical practice and clinical trials to assess disease symptoms in both children and adults. Participants respond to 7 items, including dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping, each scored on a 5-point scale based on frequency over the previous week: 0 = no days, 1 = 1 to 2 days, 2 = 3 to 4 days, 3 = 5 to 6 days, and 4 = all days. Item scores (0 to 4) are added to provide a total score range of 0 to 28. The total score reflects disease-related morbidity, and differentiates between "clear/almost clear" (0-2 points), "mild" (3-7 points), "moderate" (8-16 points), "severe" (17-24 points) and "very severe" (25-28 points) AD. A change in POEM score of 3.4 points is considered the MCID.
Percentage of Participants with a baseline POEM score ≥ 4 achieving an improvement (reduction) in POEM ≥ 4 at Month 4 | Up to 4 Months
  The POEM is a 7-item, validated questionnaire used in clinical practice and clinical trials to assess disease symptoms in both children and adults. Participants respond to 7 items, including dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping, each scored on a 5-point scale based on frequency over the previous week: 0 = no days, 1 = 1 to 2 days, 2 = 3 to 4 days, 3 = 5 to 6 days, and 4 = all days. Item scores (0 to 4) are added to provide a total score range of 0 to 28. The total score reflects disease-related morbidity, and differentiates between "clear/almost clear" (0-2 points), "mild" (3-7 points), "moderate" (8-16 points), "severe" (17-24 points) and "very severe" (25-28 points) AD. A change in POEM score of 3.4 points is considered the MCID.
Percentage of Participants achieving a POEM score of ≤2 among participants with POEM >2 at baseline | Up to 4 Months
  The POEM is a 7-item, validated questionnaire used in clinical practice and clinical trials to assess disease symptoms in both children and adults. Participants respond to 7 items, including dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping, each scored on a 5-point scale based on frequency over the previous week: 0 = no days, 1 = 1 to 2 days, 2 = 3 to 4 days, 3 = 5 to 6 days, and 4 = all days. Item scores (0 to 4) are added to provide a total score range of 0 to 28. The total score reflects disease-related morbidity, and differentiates between "clear/almost clear" (0-2 points), "mild" (3-7 points), "moderate" (8-16 points), "severe" (17-24 points) and "very severe" (25-28 points) AD. A change in POEM score of 3.4 points is considered the MCID.
Percent change in Body surface area (BSA) score from baseline | Up to 4 Months
  The investigator selects the participant's right or left hand as the measuring device. For purposes of clinical estimation, the total surface of the palm plus five digits is assumed to be approximately equivalent to 1%. Measurement of the total area of involvement by the investigator is aided by imagining if scattered plaques were moved so that they were next to each other and then estimating the total area involved. Published score bands: 0% (clear), 0.1-15.9% (mild), 16.0-39.9% (moderate), 40-100% (severe).
Mean change in BSA score from baseline | Up to 4 Months
  The investigator selects the participant's right or left hand as the measuring device. For purposes of clinical estimation, the total surface of the palm plus five digits is assumed to be approximately equivalent to 1%. Measurement of the total area of involvement by the investigator is aided by imagining if scattered plaques were moved so that they were next to each other and then estimating the total area involved. Published score bands: 0% (clear), 0.1-15.9% (mild), 16.0-39.9% (moderate), 40-100% (severe).
Percentage of Participants who are "Very much improved" or "Much improved" on the Patient Global Impression of Change (PGIC) | Up to 4 Months
  The PGIC ask participants to rate the overall change in their AD symptoms using a 7-point response scale: 1 = Very much improved, 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Minimally worse, 6 = Much worse, 7 = Very much worse. PGIC score ranges from 1 to 7 with lower score desirable.
Percentage of Participants who report symptoms to be "Minimal" or "Absent" on the Patient Global Impression of Severity (PGIS) | Up to 4 Months
  The PGIS ask participants to describe the severity of their AD symptoms at the present time using a 7-point response scale: 0= Absent, 1 = Minimal, 2 = Mild, 3 = Moderate, 4= Moderately Severe, 5 = Severe, 6 = Very Severe.
Percentage of Participants who report symptoms to be "Very satisfied" or "Extremely satisfied" on the Patient Global Impression of Treatment (PGIT) | Up to 4 Months
  PGIT-AD is a single item participant self-administered instrument designed to assess participant satisfaction or dissatisfaction with their current treatment for atopic dermatitis based on the following question: "Overall, how satisfied or dissatisfied are you with your current treatment for atopic dermatitis?". Response options range from 1 (extremely dissatisfied) to 7 (extremely satisfied).
Number of participants who used concomitant AD medications along with upadacitinib since last visit | Up to 4 Months
  Number of participants who used concomitant AD medications since last visit.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (25):
- Canada (25):
  - Dermatology Research Institute - Blackfoot Trail /ID# 246344, Calgary, Alberta
  - Laser Rejuvenation Clinics Inc. /ID# 255303, Calgary, Alberta
  - Rejuvenation Dermatology Clinic Calgary North /ID# 255623, Calgary, Alberta
  - Rejuvenation Dermatology - Edmonton Downtown /ID# 246298, Edmonton, Alberta
  - Stratica Medical /ID# 254940, Edmonton, Alberta
  - Rejuvaderm /ID# 255850, Edmonton, Alberta
  - Alpha Clinic Research Inc. /ID# 248015, Edmonton, Alberta
  - Dr. Chih-ho Hong Medical Inc. /ID# 246841, Surrey, British Columbia
  - Nova Scotia Health /ID# 248136, Halifax, Nova Scotia
  - Fiona Lovegrove Medicine Professional Corporation /ID# 255784, London, Ontario
  - Lynde Institute for Dermatology /ID# 246341, Markham, Ontario
  - Allergy Research Canada Inc. /ID# 251916, Niagara Falls, Ontario
  - SKiN Centre for Dermatology /ID# 246291, Peterborough, Ontario
  - York Dermatology Clinic and Research Centre /ID# 246921, Richmond Hill, Ontario
  - Canadian Dermatology Centre /ID# 246334, Toronto, Ontario
  - FACET Dermatology /ID# 254914, Toronto, Ontario
  - AvantDerm, Toronto, CA /ID# 250941, Toronto, Ontario
  - Evidence based medical educator Inc. /ID# 246687, Toronto, Ontario
  - Dr. Isabelle Delorme Inc. /ID# 246296, Drummondville, Quebec
  - Clinique D /ID# 247330, Laval, Quebec
  - Roula Rassi MD Inc /ID# 252563, Laval, Quebec
  - Diex Recherche Québec Inc. /ID# 247696, Québec, Quebec
  - Centre de Recherche St-Louis /ID# 252223, Québec, Quebec
  - Dre Angelique Gagne-Henley M.D. inc. /ID# 246457, Saint-Jérôme, Quebec
  - Sima Recherche inc. /ID# 248338, Verdun, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Clinical Study Report Synopsis — https://www.abbvieclinicaltrials.com/study/?id=P23-106#additional-resources-section